CLINICAL TRIAL: NCT02888938
Title: Performance of Pelvic Radiograph, CT -Scan and MRI of the Sacroiliac Joints to Diagnose Structural Sacroiliitis in a Large Cohort of Patients With Suspicion of Spondyloarthritis
Brief Title: Diagnosis of Structural Sacroiliitis in Patients With Suspicion of Spondyloarthritis (EchoSPA)
Acronym: Passerelle
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014/PasserelleEchoSPA-Loeuill
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Structural Sacro-iliitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients suspected of SpA
  Interventions: Other: pelvic radiography; Other: pelvic MRI; Other: pelvic CT-scan

INTERVENTIONS:
Other: pelvic radiography
Other: pelvic MRI
Other: pelvic CT-scan

SUMMARY:
The aims of this study are: 1° to assess the value of pelvic radiography and sacro-iliac joint (SIJ) MRI compared to CT scan of SIJ for the diagnosis of structural sacro-iliitis and 2° to quantify structural elementary lesions on MRI and for the first time on CT-scan according to a SPARCC approach in a cohort of patients with a suspicion of spondyloarthritis (ECHOSpA).

DETAILED DESCRIPTION:
Among the 489 patients of the cohort, MRI and CT examination of SIJ were performed simultaneously with pelvic radiographs in 173 patients. After harmonization, readers will be tested for inter-reader reproducibility for modified New York criteria, and scoring of each structural elementary lesion depicted on MRI (erosions, fat metaplasia, backfill, sclerosis and ankylosis) and on CT-scan (erosion, joint space narrowing, sclerosis and ankylosis). When acceptable inter-reader reproducibility will be obtained, exams will be blindly and independently scored by 2 readers (rheumatologist and/or radiologist) in the following order: 1/ pelvic radiographs, 2/ MRI, 3/ CT-scan. In case of discordance between readers for the diagnosis of sacroiliitis, an adjudicator will define the final diagnosis for each imaging method (senior rheumatologist or radiologist). Severity of each structural lesion will be scored quantitatively according to structural SPARCC approach. Only lesions observed in the synovial part of the SIJ on 2 successive slices will be taken into account.

Sensibility, specificity and concordance for the diagnosis of structural sacroiliitis for radiograph and MRI will be calculated with the CT-scan considered as the gold standard. Quantitative MRI and CT scores will be compared for each lesion: erosion, sclerosis and ankylosis. This quantitative approach will be used to explain cases of discordance or concordance for radiograph and MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected spondyloarthritis

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 173 patients issues from ECHOSpA cohort with pelvic radiograph, CT-scan and MRI of SIJ.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value of pelvic radiograph compared to CT-scan of sacro-iliac joint for the diagnosis of structural sacroiliitis | baseline
  according to New York criteria; CT-scan considered as the gold standard
Diagnostic value of MRI of sacro-iliac joint compared to CT-scan of sacro-iliac joint for the diagnosis of structural sacroiliitis | baseline
  according to New York criteria; CT-scan considered as the gold standard
Quantitative assessment of structural lesions of sacro-iliac joints on CT-scan according to SPARCC for structural assessment and adapted for CT-scan | baseline
Quantitative assessment of structural lesions of sacro-iliac joints on MRI according to SPARCC | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Damien Loeuille, Pr, Principal Investigator — Service deRhumatologie - CHRU Brabois
Locations (1):
- Service deRhumatologie - CHRU Brabois, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No